CLINICAL TRIAL: NCT06811818
Title: Comparison of Masticatory Performance of Bilateral Balanced Occlusion and Lingualized Occlusion in Complete Denture Patients
Brief Title: Masticatory Performance in Bilateral Balanced Occlusion and Lingualized Occlusion in Complete Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Seema Khattak, Dr. Seema Khattak , Principal Investigator and Resident Prosthodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: masticatory performance
Record Dates: First submitted 2025-01-19; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Masticatory Performance
Keywords: Masticatory performance , Bilateral balanced occlusion , Lingualized occlusion
MeSH Terms: interventions — Denture, Complete

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- complete denture with bilateral balanced occlusion (Active Comparator): complete denture with bilateral balanced occlusion
  Interventions: Other: complete denture with bilateral balanced occlusion
- complete denture with lingualized occlusion (Active Comparator): complete denture with lingualized occlusion
  Interventions: Other: complete denture with lingualized occlusion

INTERVENTIONS:
Other: complete denture with bilateral balanced occlusion — Participants in this group will be given complete dentures with bilateral balanced occlusion
  Arms: complete denture with bilateral balanced occlusion
Other: complete denture with lingualized occlusion — Participants in this group will be given complete dentures with lingualized occlusion
  Arms: complete denture with lingualized occlusion

SUMMARY:
This is a randomized control trial to compare masticatory performance in complete dentures with bilateral balanced occlusion or lingualized occlusion.

DETAILED DESCRIPTION:
This study is a randomized control trial to compare the masticatory efficiency of complete dentures with bilateral balanced occlusion with that of lingualized occlusion . Grouping of participants was carried out. Participants divided into two groups one receiving complete dentures with bilateral balanced occlusion and the other group receiving complete dentures with lingualized occlusion . Each participant provided with 15g of peanuts and instructed to chew until ready to swallow . The chew material than spat into the designated container and participants asked to rinse their mouth with water , with the rinse being collected in the same container . The collected material than sieved through 10-Mesh sieve followed by drying the sieved content on blotting paper for 30 minutes. The dried material subsequently weight with an electric balance with precision of 0.01 grams . Masticatory efficiency assessed through mean weight of chewed peanuts.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 45-65 years.
2. Both genders included.
3. Edentulous patients requiring complete denture.
4. Patients willing to participate in the study .

Exclusion Criteria:

1. Participants not willing to participate in the study.
2. Participants with systemic disease .
3. Participants with neuromuscular disorders .

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Masticatory Efficiency in Complete Dentures by weighing the dried chewed material through electric balance | upto 24 weeks
  The chewed material that has been sieved through 10-mesh sieve and dried through blotting paper for 30 minutes weighted using an electronic balance with a precision of 0.01 grams . Statistical analysis performed to evaluate masticatory efficiency based on the mean weight of chewed peanuts.

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khattak, BDS, Principal Investigator — Armed Forces Institute of Dentistry
Locations (1):
- Armed Forces Institute Of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No